CLINICAL TRIAL: NCT03154099
Title: Critical Illness Related Corticosteroid Insufficiency
Brief Title: Critical Illness Related Corticosteroids Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma mohammad, Assiut, Assiut University
Other Study IDs: assiut univeristy13577
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2017-05

CONDITIONS: Prevalence of CIRCI . Most Common Presentations of CIRCI . the Best Method of Replacment
Keywords: CIRCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the detrimental impact of dysfunction is well recognized. CIRCI may be characterized by any of the following findings with delayed weaning from mechanical ventilation and hypotension refractory to fluids and vasopressors being most common Hypotension Unresponsiveness to catecholamine infusions Ventilator dependence Abdominal or flank pain High fever with negative cultures and unresponsive to antibiotic therapy Unexplained mental changes (i.e., apathy or depression) Electrolyte abnormalities (hypoglycemia, hyponatremia, hyperkalemia) Neutropenia, eosinophilia

DETAILED DESCRIPTION:
Critically ill patients are at risk for the development of Critical Illness-Related Corticosteroid Insufficiency (CIRCI). This may present as hypotension, unresponsiveness to catecholamine infusions, and/or ventilator dependence. Such patients may benefit from administration of exogenous steroids to restore their hemodynamic stability. Cortisol is vitally important to the maintenance of vascular tone, endothelial integrity, vascular permeability, and total body water distribution. It also potentiates the vasoconstrictor actions of both endogenous and exogenous catecholamines. Appropriate activation of the hypothalamic-pituitary-adrenal (HPA) axis in the critically ill patient is essential to stress adaptation and maintenance of homeostasis. Common causes of adrenal insufficiency in the critical care setting include infection, systemic inflammation, previous glucocorticoid use, and sepsis . Adrenal insufficiency among critically ill patients is also known as relative adrenal insufficiency; there is either insufficient cortisol or a cortisol level that may be high in absolute terms but insufficient to respond to the degree of stress. Thus, serum cortisol concentrations that are normal in well patients may be inappropriately low in severely sick patients. This inability to mount the appropriate response increases the risk of death during severe illness. While the incidence of CIRCI in the critically ill has been under appreciated, the detrimental impact of such dysfunction is well recognized. CIRCI may be characterized by any of the following findings with delayed weaning from mechanical ventilation and hypotension refractory to fluids and vasopressors being most common Hypotension Unresponsiveness to catecholamine infusions Ventilator dependence Abdominal or flank pain High fever with negative cultures and unresponsive to antibiotic therapy Unexplained mental changes (i.e., apathy or depression) Electrolyte abnormalities (hypoglycemia, hyponatremia, hyperkalemia) Neutropenia, eosinophilia Diagnostic criteria for CIRCI in the critically ill are not well established, but evidence suggests that modifications from standard testing are warranted. Random serum cortisol levels, free cortisol, and delta cortisol (change in baseline cortisol at 60 minutes after ACTH stimulation using 250 mcg cosyntropin) are all ways to evaluate for CIRCI.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit all critically ill patients in Critical Care Unit with APACHE II score >25.

Exclusion Criteria:

* A known patient with adrenal insufficiency.
* Patient with a previous history of steroid therapy for more than one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit all critically ill patients >18 years in Critical Care Unit with APACHE II score >25 then we mesure Random serum cortisol levels and delta cortisol (change in baseline cortisol at 60 minutes after ACTH stimulation using 250 mcg cosyntropin) are all ways to evaluate for CIRCI
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Critical illness related corticosteroid insufficiency | one year
  Prevalence of CIRCI . most common presentations of CIRCI . the best method of replacment we mesure Random serum cortisol levels and delta cortisol (change in baseline cortisol at 60 minutes after ACTH stimulation using 250 mcg cosyntropin) are all ways to evaluate for CIRCI.

IPD SHARING:
Plan to Share IPD: Undecided
Prevalence of CIRCI . most common presentations of CIRCI . the best method of replacment